CLINICAL TRIAL: NCT01142921
Title: A Prospective Randomised Study on the Patency Period of the Plastic Anti-reflux Biliary Stent
Brief Title: The Patency Period of the New Plastic Anti-reflux Biliary Stent
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Issue regarding the stent design
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARBS
Record Dates: First submitted 2010-06-08; First posted 2010-06-14 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Pancreatitis; Cholangitis
Keywords: Stent Occlusion; Biliary Bleeding; Biliary Perforation
MeSH Terms: conditions — Pancreatitis; Cholangitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ordinary Tannenbaum biliary stent (Active Comparator): Ordinary Tannenbaum biliary stent
  Interventions: Device: Ordinary Tannenbaum biliary stent
- Anti-reflux Tannenbaum biliary stent (Experimental): Anti-reflux Tannenbaum biliary stent
  Interventions: Device: Anti-reflux Tannenbaum biliary stent

INTERVENTIONS:
Device: Anti-reflux Tannenbaum biliary stent — Anti-reflux Tannenbaum biliary stent
  Other Names: Fusion® Marathon™ Anti-Reflux Biliary Stent
  Arms: Anti-reflux Tannenbaum biliary stent
Device: Ordinary Tannenbaum biliary stent — Ordinary Tannenbaum biliary stent
  Other Names: ST-2 Soehendra® Tannenbaum® Biliary Stent
  Arms: Ordinary Tannenbaum biliary stent

SUMMARY:
The aim of this study is to determine the average patency period of the new anti-reflux biliary stent on patients with malignant bile duct strictures and to determine if this stent remains patent for a longer period of time comparing with the ordinary plastic Tannenbaum biliary stent.

DETAILED DESCRIPTION:
Bile duct related cancer is a condition quite commonly seen among Asians. Predisposing conditions for primary bile duct cancer include recurrent infections and autoimmune diseases such as recurrent pyogenic cholangitis (RPC) and primary sclerosing cholangitis (PSC) as well as congenital problem such as choledochal cyst. Peri-ampullary tumour, pancreatic tumour and metastatic tumours with bile duct compression are other causes of bile duct obstruction. As many of these tumours are discovered at a late stage, curative treatment is usually not feasible. Palliative endoscopic stenting of the obstructed biliary system remains the treatment of choice for the majority.

The main problem with endoscopic stenting of the biliary system is the short stent patency period. There are some reports on modifications to plastic biliary stenting method in recent years including changes in stent designs, use of a different material or coating, administrating prophylactic antibiotics and the use of special drugs. All these have failed to show any conclusive effect on the stent patency period.

A preliminary study has demonstrated some promising results in the use of a stent with an anti-reflux property very similar to the stents the investigators are using in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old
* Patients who have cholangiographic evidence (on ERCP) consistent with a malignant extrahepatic biliary stricture (below bifurcation of the common hepatic duct) who require plastic stenting
* Patients with peri-ampullary tumours, pancreatic tumours, gall bladder cancer and metastatic tumours with suspected extrinsic bile duct compression
* Patients with stent or nasobiliary drain in-situ without previous sphincterotomy will qualify for the study if they satisfy the above inclusion criteria.

Exclusion Criteria:

* Patients fit for surgery.
* Patients who have dominant biliary strictures involving the hilum or more proximal biliary segments.
* Previous sphincterotomy.
* Other medical conditions that will result in a life expectancy of less then 3 months (ASA class >4)
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
time-to-occlusion or stent patency period in days | within 25 weeks of device application

SECONDARY OUTCOMES:
Bleeding associated with endoscopic retrograde cholangiopancreatography (ERCP) and stent placement | within 25 weeks of device application
perforation associated with ERCP and stent placement | within 25 weeks of device application
pancreatitis associated with ERCP and stent placement | within 25 weeks of device application
cholangitis associated with ERCP and stent placement | within 25 weeks of device application
stent migration associated with ERCP and stent placement | within 25 weeks of device application
all cause mortality | within 25 weeks of device application

CONTACTS AND LOCATIONS:
Overall Officials: Wai L Quan, Dr., Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Centre, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leong QW, Shen ML, Au KW, Luo D, Lau JY, Wu JC, Chan FK, Sung JJ. A prospective, randomized study of the patency period of the plastic antireflux biliary stent: an interim analysis. Gastrointest Endosc. 2016 Feb;83(2):387-93. doi: 10.1016/j.gie.2015.04.027. Epub 2015 May 27. PMID 26024583